CLINICAL TRIAL: NCT06468475
Title: Enhancing Neonatal Sucking Reflex: A Study on the Efficacy of Magnesium Sulphate in Severe Birth Asphyxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RESnTEC, Institute of Research (Other)
Responsible Party: Principal Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHMULTAN
Record Dates: First submitted 2024-06-15; First posted 2024-06-21 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Birth Asphyxia
MeSH Terms: conditions — Asphyxia Neonatorum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium Sulphate Group (Experimental)
  Interventions: Drug: Magnesium Sulphate infusion
- Control (No Intervention)

INTERVENTIONS:
Drug: Magnesium Sulphate infusion — Magnesium sulphate 24 hours apart by intravenous infusion at 250 mg/kg/dose (0.5 mL/kg/dose of injection magnesium sulphate 50% w/v diluted in 5 mL/kg of 5% glucose) over a duration of half an hour by an infusion pump
  Arms: Magnesium Sulphate Group

SUMMARY:
Children's Hospital Multan is a tertiary care teaching hospital in South Punjab, the poorest and most backward area of Punjab, Pakistan, where a significant number of newborns suffer from birth asphyxia. Therefore, this study was planned with the objective of investigating the effectiveness of magnesium sulphate in severe birth asphyxia, hypothesizing that in cases of birth asphyxia, neonates who are treated with magnesium sulphate have a higher sucking reflex than those who are not treated with magnesium sulphate.

ELIGIBILITY:
Inclusion Criteria:

* Full-term babies (≥37 weeks of gestation)
* Both genders
* Severe birth asphyxia
* Admitted within six hours of life.

Exclusion Criteria:

* Premature babies
* Congenital malformations
* Babies born to mothers who received general anesthesia
* Babies whose mothers received magnesium sulfate, pethidine, and other drugs in the past 7 days.

Ages: 1 Hour to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Efficacy | 72 hours
  Efficacy was labeled as yes if the infant was placed in the supine position, the index finger was placed in the infant's mouth, and the power of sucking movements was judged after 5 seconds, and If the sucking reflex appeared. Efficacy was termed no otherwise.

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital and the Institute of Child Health, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared with researchers on a reasonable request